CLINICAL TRIAL: NCT06958575
Title: Outcomes Assessment of Septal Extension Graft Versus Columellar Strut Graft in Rhinoplasty.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hossam Aldein Samir Abd Elazeem Mohammed, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: septal extension graf
Record Dates: First submitted 2025-04-14; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Septal Extension Graft in Rhinoplasty
Keywords: Rhinoplasty; Septal extension graft

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Septal extension graft will be used. The triangle-shaped cartilage graft prepared from the septal cartilage is placed into one or bothsides of the caudal septum reciprocally according to its structure and curvature and sutured with horizontal mattress sutures. After graft stabilization, two insulin needles are passed through the medial crura and the graft to determine its level of placement. After the rotation and nasal projection are adjusted, the medial crura are sutured to the septal extension grafts.
  Interventions: Procedure: Septal extension graft
- Group 2 (Active Comparator): Columellar strut graft will be used. A strut graft 10-12 mm long is placed into a web created between the two medial crura and stabilized by sutures placed between the graft and medial crura.
  Interventions: Procedure: Columellar strut

INTERVENTIONS:
Procedure: Septal extension graft — Septal extension graft will be used. The triangle-shaped cartilage graft prepared from the septal cartilage is placed into one or bothsides of the caudal septum reciprocally according to its structure and curvature and sutured with horizontal mattress sutures. After graft stabilization, two insulin needles are passed through the medial crura and the graft to determine its level of placement. After the rotation and nasal projection are adjusted, the medial crura are sutured to the septal graft.
  Arms: Group 1
Procedure: Columellar strut — Columellar strut graft will be used. A strut graft 1012 mm long is placed into a web created between the two medial crura and stabilized by sutures placed between the graft and medial crura.
  Arms: Group 2

SUMMARY:
Nose is an important aesthetic landmark with its length, width, shape, and position in the middle of the face. Rhinoplasty is now one of the most common rhinological procedures with both functional and aesthetic aspects. Tip plasty is considered the core of rhinoplasty. The interaction among lower lateral cartilages, septal cartilage, adjacent soft tissues, tissue dynamics, and surgical techniques determines the nasal tips projection, rotation, and overall shape. Various graft sources and types were used for tip support in rhinoplasty such as columellar struts, septal extensions, and cap grafts.

The columellar strut graft, first introduced in 1932, has became a widely adopted technique. Typically a cartilage graft is positioned between the medial crura to provide support and stability to the nasal tip. Recent studies reported some drawbacks of columellar strut such as widening the columella and resorption or displacement of the graft due to their lack of attachment to the caudal septum. Septal extension grafts extend from the caudal edge of the nasal septum into the lower lateral cartilages, these grafts offer crucial structural support to the nasal tip. Despite of their the wide use of columellar strut and septal extention graft, limited studies compared their results.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (more than 18 years).
2. Patients with any type of tip deformaties.
3. Patients fit for surgery.

Exclusion Criteria:

1. Patients with history of previous nasal surgery.
2. Pregnant patients.
3. Patients with chronic diseases affecting wound healing e.g. DM and blood diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Tip projection and rotation | These values will be evaluated before surgical intervention and 6 months after the surgery
  Two factors will be assessed to compare the changes of tip projection and rotation in each group: the ratio of nasal projection to nasal length and the columellar-labial angle values.
  The program Rhinobase developed by Apaydin et Al. will be used for photographic analysis to calculate the the ratio of nasal projection to nasal length and the columella labial angle values. This software allowed for consistent and objective measurements that were independent of the individual performing the analysis, minimizing variability. These values will be evaluated before surgical intervention and 6 months after the surgery.

SECONDARY OUTCOMES:
Patient satisfaction | Before and 6 months after the surgery.
  Patient satisfaction will be assessed using an arabic version of validated rhinoplasty outcome evaluation (ROE) questionnaire six months after the surgery. The questionnaire is consist of six questions and each question is scored on 0-4 scale:
  0: worest possible outcome. 4:best possible outcome. The score from the six questions are summed up to give the total score. The total is then divided by 24 (the maximum score) and multiplied by 100 to get a percentage.

IPD SHARING:
Plan to Share IPD: Undecided